CLINICAL TRIAL: NCT06849596
Title: A Cluster Crossover Randomized Controlled Trial of Manual T-piece Versus Ventilator Positive Pressure Ventilation During Resuscitation of Extremely Premature Neonates: The MVP Trial
Brief Title: Manual T-piece Versus Ventilator Positive Pressure Ventilation During Resuscitation of Extremely Premature Neonates
Acronym: MVP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Baczynski (Other)
Collaborators: Royal Alexandra Hospital (Other); Foothills Medical Centre (Other); McMaster Children's Hospital (Other); St. Justine's Hospital (Other); Cedars-Sinai Medical Center (Other); Montreal Children's Hospital of the MUHC (Other); Sunnybrook Health Sciences Centre (Other); London Health Sciences Centre (Other); BC Women's Hospital & Health Centre (Other)
Responsible Party: Sponsor-Investigator, Michelle Baczynski, Respiratory Therapist, Mount Sinai Hospital, Canada
Organization: Mount Sinai Hospital, Canada (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CTO 5018
Record Dates: First submitted 2024-12-13; First posted 2025-02-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Resuscitation; Apnea Neonatal
Keywords: Premature Infant; Preterm Neonates; Oxygen; Lung Injury; Respiration, Artificial; Resuscitation; Ventilator, Mechanical
MeSH Terms: conditions — Premature Birth; Lung Injury; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: This study will be a cluster-crossover, unmasked randomized control trial (RCT) comparing the clinical effectiveness of two existing methods for providing PPV to preterm neonates born 25+0 to 28+6 weeks gestational age during initial resuscitation after birth.
Who Masked: Outcomes Assessor
Masking Description: The DSMB will assess intervention compliance and mortality rates, masked to the group allocation. The trial statistician will be blinded to group allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (T-Piece Resuscitator) (Active Comparator): Positive pressure ventilation during the first 10 minutes after birth will be provided with a T-Piece Resuscitator (TPR; Neopuff, Fisher & Paykel Healthcare) connected to an appropriately sized face-mask, with settings adjustable within specified ranges for positive inspiratory pressure, positive end expiratory pressure, and fraction of inspired oxygen based on local policy. These specified ranges will be standardized across sites.
  Interventions: Device: T-piece resuscitator (TPR)
- Intervention under investigation (Ventilator delivered PPV) (Experimental): Positive pressure ventilation (PPV) during the first 10 minutes after birth will be provided using a neonatal ventilator set up in noninvasive positive pressure ventilation (NIPPV) mode, connected to an appropriately sized nasal mask or prongs and a dual limb neonatal ventilator circuit, with settings adjustable within specified ranges for positive inspiratory pressure, positive end expiratory pressure, respiratory rate and inspiratory time and fraction of inspired oxygen based on local policy. These specified ranges will be standardized across sites.
  Interventions: Device: Ventilator derived positive pressure ventilation - V-PPV

INTERVENTIONS:
Device: Ventilator derived positive pressure ventilation - V-PPV — The clinical team will determine the need for PPV, as per local practice and Neonatal Resuscitation Program. Each site will be previously randomized to their method of providing PPV for preterm neonates during the first 10 minutes after birth. Ventilator delivered positive pressure ventilation (V-PPV) using a nasal interface will be delivered to the infant in the resuscitation room.
  Arms: Intervention under investigation (Ventilator delivered PPV)
Device: T-piece resuscitator (TPR) — The clinical team will determine the need for PPV, as per local practice and Neonatal Resuscitation Program. Each site will be previously randomized to their method of providing PPV for preterm neonates during the first 10 minutes after birth. PPV will be provided with a T-piece resuscitator (Neopuff, Fisher & Paykel Healthcare) connected to an appropriately sized face-mask.
  Arms: Control group (T-Piece Resuscitator)

SUMMARY:
Many extremely premature infants require immediate help with breathing after birth. Positive pressure ventilation (PPV) using a device called a T-piece resuscitator is a common method. PPV is needed to establish proper lung function, improve gas exchange, and encourage the infant to breathe spontaneously. However, T-piece resuscitators have limitations, like a lack of visual feedback and variable settings, which may result in reduced effectiveness of PPV. Improving PPV effectiveness may reduce the need for more invasive procedures, such as intubation, which pose an increased risk of complications and death for these fragile infants. A novel approach, that may overcome the above limitations and deliver PPV with precise settings through a nasal mask, is to use a ventilator to deliver PPV (V-PPV) using a respiratory mode called nasal intermittent positive pressure ventilation (NIPPV). While NIPPV is commonly used in neonatal intensive care units to support breathing in premature infants, the impact of V-PPV use during immediate post-birth stabilization needs to be studied. Preliminary data from our recent single-center study confirmed the feasibility of using V-PPV for resuscitation of extremely premature babies and indicated its potential superiority with a 28% decrease in the need for intubation compared to historical use of T-piece. This promising innovation may enhance outcomes for these vulnerable infants by refining the way we provide respiratory support in their critical first moments. The research objective is to compare the clinical outcomes of extremely premature infants receiving manual T-piece versus V-PPV during immediate post-birth stabilization. The primary aim is to evaluate the impact of V-PPV on major health complications or death. This study seeks to provide insights into improving the care and outcomes of these infants during a critical stage of transition from fetus to newborn.

ELIGIBILITY:
Inclusion Criteria::

* GA 25+0 to 28+6 weeks using the best available obstetrical estimate
* Designated to receive full resuscitation, i.e., not pre-determined to receive only comfort care
* Received PPV as determined by the resuscitation team during the first 10 minutes of birth

Exclusion Criteria:

* Outborn birth status
* Resuscitation performed in unforeseen circumstances outside typical delivery room (e.g., emergency department, antenatal ward)
* Known major congenital or chromosomal anomaly
* Established spontaneous respiration without receipt of PPV

Ages: 25 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 780 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite of pre-discharge mortality | From enrollment through study completion (up to 50 weeks postmenstrual age)
  Death in NICU
Major neuro-injury | From enrollment through study completion (up to 50 weeks postmenstrual age)
  Defined as IVH ≥grade 3, cerebellar hemorrhage or periventricular leukomalacia.
Moderate-severe BPD | At 36 weeks' postmenstrual age.
  Defined as 2 L/min nasal cannula or other forms of non-invasive ventilation support or invasive mechanical ventilation.

SECONDARY OUTCOMES:
Components of the primary outcome | From enrollment through study completion (up to 50 weeks postmenstrual age)
  Pre-discharge mortality, major neuro-injury or moderate-severe BPD
Frequency of receipt of advanced cardiopulmonary resuscitation measures | From enrollment to 1 hour post intervention.
  Chest compressions or epinephrine administration for the purpose of resuscitation.
Duration of invasive mechanical ventilation during NICU admission | From enrollment through study completion (up to 50 weeks postmenstrual age)
  Total number of days on invasive mechanical ventilation
Discharge on home oxygen | From enrollment through study completion (up to 50 weeks postmenstrual age)
  Discharge from the NICU requiring oxygen support at home
Other relevant key prematurity related adverse outcome | From enrollment through study completion (up to 50 weeks postmenstrual age)
  Necrotizing enterocolitis ≥ stage 2a, retinopathy of prematurity needing treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Baczynski, MSc, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (10):
- Cedars-Sinai Guerin Children's, Los Angeles, California, United States
- Canada (8):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - BC Children's and Women's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital at London Health Sciences Centre, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Montreal Children's Hospital, Montral, Quebec
  - CHU Sainte Justine, Montreal, Quebec
- Rigshospitalet Coppenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No